CLINICAL TRIAL: NCT02581449
Title: Evaluation of the Effect of Omega-3 Fatty Acids Supplementation on Pediatric Patients Undergoing Hemodialysis
Brief Title: Effect of Omega-3 Fatty Acids on Oxidative Stress and Dyslipidemia in Pediatric Patients Undergoing Hemodialysis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Areej Mohamed Ateya, teaching assistant, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PHCL31528
Record Dates: First submitted 2015-10-11; First posted 2015-10-21 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: End Stage Renal Disease
Keywords: omega-3 fatty acids; hemodialysis; oxidative stress; dyslipidemia
MeSH Terms: conditions — Kidney Failure, Chronic; Dyslipidemias | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- omega-3 group (Experimental): omega-3 soft gelatin capsules 1000 mg (500mg EPA+250mg DHA)once daily for four months
  Interventions: Dietary Supplement: omega-3
- placebo group (Placebo Comparator): empty soft gelatin capsules with matched size, color and shape once daily for four months
  Interventions: Other: empty soft gelatin capsules

INTERVENTIONS:
Dietary Supplement: omega-3 — dietary supplement
  Other Names: NOW foods omega-3 softgels
  Arms: omega-3 group
Other: empty soft gelatin capsules — empty softgels of matched size, shape and color
  Arms: placebo group

SUMMARY:
The purpose of the study is to evaluate the effect of omega-3 fatty acids supplementation on pediatric patients undergoing hemodialysis via the measurement of the following before and after omega-3 administration:oxidative stress markers, inflammatory markers and serum lipids.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 8 and 18 years old
* Patients treated with HD for at least 6 months

Exclusion Criteria:

* Patients with malignancy and active inflammatory disease.
* Patients who received vitamin E or any antioxidant treatment during the past 3 months.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-09; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
effect on oxidative stress status via measurement of superoxide dismutase and glutathione peroxidase and malondialdehyde | four months

SECONDARY OUTCOMES:
effect on serum lipid levels (HDL cholesterol, LDL cholesterol, total cholesterol, and triglycerides) | four months

OTHER OUTCOMES:
effect on inflammation via measurement of C- Reactive Protein | four months
effect on nitric oxide (serum concentration) | four months

CONTACTS AND LOCATIONS:
Overall Officials: Ain Shams, Principal Investigator — university